CLINICAL TRIAL: NCT06700408
Title: Efficacy and Safety of Dachaihu Decoction Combined Erzhiwan With Variation for the Treatment of Hypercholesterolemia: A Parallel, Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: RCT for the Chinese Medicine in Treating Hypercholesterolemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Hypercholesterolemia study
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dachaihu Decoction combined Erzhiwan with variation granules (Experimental): Chinese medicine granules
  Interventions: Drug: Dachaihu Decoction combined Erzhiwan with variation
- Placebo granules (Placebo Comparator): Placebo granules
  Interventions: Other: Placebo granules

INTERVENTIONS:
Drug: Dachaihu Decoction combined Erzhiwan with variation — Chinese medicine granules
  Other Names: Chinese medicine granules
  Arms: Dachaihu Decoction combined Erzhiwan with variation granules
Other: Placebo granules — Placebo granules
  Arms: Placebo granules

SUMMARY:
This is a randomized, double-blind, placebo-controlled clinical trial. Eligible subjects will randomized into a treatment group or placebo group. They will receive either Chinese medicine granules or placebo granules for 8 weeks followed by a 4-week observation period. The primary outcome would be the percent change in Low-density lipoprotein cholesterol levels (LDL-C) after treatment.

DETAILED DESCRIPTION:
Hypercholesterolemia refers to a metabolic disease caused by abnormal cholesterol metabolism in the blood cholesterol content exceeding the normal range, which can be mainly divided into total cholesterol (TC) in plasma and low-density lipoprotein cholesterol LDL-C) or a decrease in high-density lipoprotein cholesterol (HDL-C). Uncontrolled hypercholesterolemia is considered an important risk factor for cardiovascular and cerebrovascular diseases.

In recent years, there has been an increasing number of clinical studies of Traditional Chinese Medicine combinations or single herbs for hypercholesterolemia, and some drugs do have cholesterol-lowering effects, but the clinical evidence is not high due to bias or other deficiencies in trial design. Therefore, this clinical trial aim to evaluate the effectiveness of Dachaihu Decoction combined Erzhiwan with variation to the treatment of patients with clinical hypercholesterolemia, and tried to reduce its adverse effects on liver function through reasonable compatibility.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years old, any gender;
* LDL-C level of 4.1 mmol/L or above (no statin therapy during the screening period);
* Be able to maintain a more consistent lifestyle and eating habits throughout the study;
* Have a fixed residence and are not expected to move or travel for 8 weeks;
* Voluntarily sign the informed consent form.

Exclusion Criteria:

* Taking drugs that may affect lipid metabolism (such as steroids, sleeping pills, and psychotropic drugs);
* Alcohol or drug abuse within the last 3 months;
* Known liver function or renal dysfunction;
* History of severe cardiovascular and cerebrovascular diseases; or history of psychiatric illness;
* Participate in other interventional clinical trials within 3 months before the study, including drugs, supplements, medical devices, etc.;
* Known pregnant or lactating women, allergies or allergies to traditional Chinese medicine;
* Patients with known secondary hypercholesterolemia.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
The percent change in Low-density lipoprotein-cholesterol (LDL-C) levels | 8 weeks
  Compare the percent change in LDL-C levels from baseline to week 8

SECONDARY OUTCOMES:
The percent change in Low-density lipoprotein-cholesterol (LDL-C) levels | 4 weeks
  Compare the percent change in LDL-C levels from baseline to week 4
The percent change in Low-density lipoprotein-cholesterol (LDL-C) levels | 12 weeks
  Compare the percent change in LDL-C levels from baseline to week 12
The level of Low-density lipoprotein-cholesterol (LDL-C) | 4 weeks
  The level of LDL-C at week 4
The level of Low-density lipoprotein-cholesterol (LDL-C) | 8 weeks
  The level of LDL-C at week 8
The level of Low-density lipoprotein-cholesterol (LDL-C) | 12 weeks
  The level of LDL-C at week 12
The percent change in High-density lipoprotein-cholesterol (HDL-C) level | 4 weeks
  Compare the percent change in HDL-C levels from baseline to week 4
The percent change in High-density lipoprotein-cholesterol (HDL-C) level | 8 weeks
  Compare the percent change in HDL-C levels from baseline to week 8
The percent change in High-density lipoprotein-cholesterol (HDL-C) level | 12 weeks
  Compare the percent change in HDL-C levels from baseline to week 12
The level of High-density lipoprotein-cholesterol (HDL-C) | 4 weeks
  The level of HDL-C at week 4
The level of High-density lipoprotein-cholesterol (HDL-C) | 8 weeks
  The level of HDL-C at week 8
The level of High-density lipoprotein-cholesterol (HDL-C) | 12 weeks
  The level of HDL-C at week 12
The percent change in Total cholesterol (TC) level | 4 weeks
  Compare the percent change in TC levels from baseline to week 4
The percent change in Total cholesterol (TC) level | 8 weeks
  Compare the percent change in TC levels from baseline to week 8
The percent change in Total cholesterol (TC) level | 12 weeks
  Compare the percent change in TC levels from baseline to week 12
The level of Total cholesterol (TC) | 4 weeks
  The level of HDL-C at week 4
The level of Total cholesterol (TC) | 8 weeks
  The level of HDL-C at week 8
The level of Total cholesterol (TC) | 12 weeks
  The level of HDL-C at week 12
The percent change in Triglycerides (TG) | 4 weeks
  Compare the percent change in TC levels from baseline to week 4
The percent change in Triglycerides (TG) | 8 weeks
  Compare the percent change in TC levels from baseline to week 8
The percent change in Triglycerides (TG) | 12 weeks
  Compare the percent change in TC levels from baseline to week 12
The level of Triglycerides (TG) | 4 weeks
  The level of Triglycerides (TG) at week 4
The level of Triglycerides (TG) | 8 weeks
  The level of Triglycerides (TG) at week 8
The level of Triglycerides (TG) | 12 weeks
  The level of Triglycerides (TG) at week 12
Proportion of patients' LDL-c below 70 mg/L | 8 weeks
  The proportion of patients in the two groups who achieved LDL-C levels below 70 mg/L at week 8
Proportion of patients' LDL-c below 70 mg/L | 12 weeks
  The proportion of patients in the two groups who achieved LDL-C levels below 70 mg/L at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, Prof, Principal Investigator — Chinese University of Hong Kong

IPD SHARING:
Plan to Share IPD: No